CLINICAL TRIAL: NCT04378842
Title: Impact of SARS-CoV-2 Infection on the Incidence of ICU Acquired Colonization Related to Multidrug-resistant Bacteria
Brief Title: COVID-19 and ICU-acquired MDR Bacteria
Acronym: COVID-BMR
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_37; 2020-A01157-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Sars-CoV2; Critical Illness
Keywords: Covid-19; Critically ill patients; multidrug-resistant bacteria; infection; colonization
MeSH Terms: conditions — Critical Illness; COVID-19; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter before-after study aimed to determine the impact of infection related to SARS-CoV-2 on the incidence of ICU-acquired multidrug resistant (MDR) bacteria.

DETAILED DESCRIPTION:
Multicenter observational before-after study, aiming to determine the impact of infection related to SARS-CoV-2 on the incidence of ICU-acquired colonization and infection related to MDR bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Expected ICU stay > 48 hours
* Rectal and nasal BMR screening performed < 48 hours after admission to ICU

Exclusion Criteria:

* Patients aged < 18 years Refusal to take part in the study ICU-stay < 48 hours At least a second rectal and nasal BMR screening was not performed prior to ICU discharge (a posteriori exclusion criterion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to intensive care
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of ICU-acquired colonization related multidrug resistant bacteria | from D3 until day 28 after ICU admission
  percentage of patients with ICU acquired MDR bacteria colonization

SECONDARY OUTCOMES:
Cumulative incidence of ICU-acquired infection related to multidrug resistant bacteria | from D3 until day 28 after ICU admission
  percentage of patients with ICU acquired MDR bacteria infection
Mechanical ventilation duration | from D1 until day 28 after ICU admission
  the number of days Under mechanical ventilation
mortality | from D1 until day 28 after ICU admission
  death in the ICU
length of stay in intensive care unit | from D1 until day 28 after ICU admission
  the number of days of hospitalization in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - Chu Amiens Picardie, Amiens
  - Ch Bethune, Béthune
  - Grand Hopital de L'Est Francilien, Jossigny
  - CH LENS, Lens
  - Hôpital Roger Salengro, ICU, CHU Lille, Lille
  - Hospices Civils de Lyon (Pierre Bénite,Edouard Herriot, La Croix Rousse), Lyon
  - Hospices Civils de Lyon, Lyon

REFERENCES:
- [Derived] Kreitmann L, Jermoumi S, Vasseur M, Chabani M, Nourry E, Richard JC, Wallet F, Garcon P, Kachmar S, Zerbib Y, Van Grunderbeeck N, Vinsonneau C, Duhamel A, Labreuche J, Nseir S. Relationship between COVID-19 and ICU-acquired colonization and infection related to multidrug-resistant bacteria: a prospective multicenter before-after study. Intensive Care Med. 2023 Jul;49(7):796-807. doi: 10.1007/s00134-023-07109-5. Epub 2023 Jun 16. PMID 37326645